CLINICAL TRIAL: NCT02992821
Title: Screening Patients Admitted With Stroke or TIA for Carotid Stenosis by Pocked-Sized Ultrasound in Inexperienced Hands and With Novel Doppler Technology
Brief Title: Pocket Sized Carotid Stenosis Screening by Junior Doctors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS_Carot_16
Record Dates: First submitted 2016-12-05; First posted 2016-12-14 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Attack, Transient; Transient Ischemic Attack; Stroke; Cerebrovascular Accident; Cerebrovascular Apoplexy
Keywords: Hand-held; Ultrasound; Diagnosis; Carotid artery stenosis
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Disease; Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bed-side pocket-size ultrasound (Experimental): All participants will be examined bed-side by pocket size ultrasound for the assessment of the carotid arteries by junior doctors. All participants will then be examined by reference imaging in specific ultrasound laboratories with conventional high end equipment and new doppler techniques and when appropriate computer tomography or magnetic resonance imaging.
  Interventions: Procedure: Bed-side pocket size ultrasound imaging; Procedure: High frame rate tracking doppler

INTERVENTIONS:
Procedure: Bed-side pocket size ultrasound imaging
  Other Names: GE Ultrasound V-scan Duo probe
Procedure: High frame rate tracking doppler
  Other Names: Verasonics research scanner

SUMMARY:
Among patients admitted with cerebral ischemia (stroke and transitory ischemic attack (TIA)) it is important to reveal the underlying cause of the disease. In special it is important to reveal if carotid artery stenosis is present as such a finding will directly influence on treatment and follow-up.

For the diagnosis of carotid artery stenosis due to atherosclerosis ultrasound examinations is the cornerstone, but computer tomography and magnetic resonance imaging may be better in some cases. Development of high quality pocket-sized ultrasound scanners has allowed for semi quantitatively bed-side assessment of the carotid arteries and the heart.

The investigators aim to study the feasibility and reliability of bed-side assessment of the carotid arteries by pocket-sized ultrasound scanners in inexperienced hands and the clinical influence of this examination when performed by experienced users.

The investigators hypothesize that a significant proportion of this patient population can be clarified bed-side by junior doctors with no need of further imaging procedures for the assessment of the carotid arteries and the heart.

DETAILED DESCRIPTION:
Population: Approximately 100 patients admitted to the Department of Medicine, Levanger Hospital and Stroke Department, St. Olavs Hospital with history and findings suspicious of stroke/transitory ischemic attack (TIA). Informed consent mandatory.

Exclusion criteria: CT angiography of carotid vessels performed after index event, unless all participating clinicians are fully blinded to the results.

Hypotheses:

The carotid arteries can be assessed bed-side by pocket-size ultrasound scanners with high feasibility and reliability by junior doctors with limited training.

Bed-side assessment of the carotid arteries by pocket-size ultrasound scanners may reduce the need for more advanced (higher cost) imaging procedures.

New high frame rate tracking doppler can increase accuracy and reproducability of stenosis grading.

Methods:

Pocket-size imaging device from GE Ultrasound, commercial available. Approved for clinical use. High-end carotid Doppler ultrasound by high-end equipment (GE Vivid 9) and computer tomography and magnetic resonance imaging at the Department of Radiology, Levanger Hospital and St. Olavs Hospital Verasonics research scanner for high fram rate imaging

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Department of Medicine with history and findings suspicious of (transient) cerebrovascular ischemia and willing and able to give their informed written consent

Exclusion Criteria:

* Evaluation of carotid artery stenosis by imaging (CT, MRI or ultrasound) performed during the stay prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without need for further diagnostic imaging | The participants will be followed for the duration of hospital stay, an expected average of approximately 4 days
  Proportion of patients which is not in need of further imaging procedures of the carotid arteries after bed-side diagnostic ultrasound performed by junior doctors with with pocket-sized scanner

SECONDARY OUTCOMES:
Reliability of bed-side ultrasound examinations of the carotid arteries performed by junior doctors with pocket-sized scanners | The participants will be followed for the duration of hospital stay, an expected average of approximately 4 days
  The accuracy of semi quantitatively classifications (like i.e. non-significant atherosclerosis of the carotid arteries vs significant stenosis of the carotid arteries) of bed-side ultrasound examinations of the carotid arteries performed by junior doctors with pocket-sized scanners compared with reference methods performed by experienced personnel
Proportion of interpretable examinations with bed-side ultrasound examinations of the carotid arteries performed by junior doctors with pocket-sized scanners | The participants will be followed for the duration of hospital stay, an expected average of approximately 4 days
  Proportion of bed-side ultrasound examinations of the carotid arteries performed by junior doctors with pocket-sized scanners of sufficient quality compared with reference imaging methods. Quality includes both to what extent the specific structure can be completely assessed, and to what degree the recordings can be interpreted by the operator. Structures and specific functions to be tested: carotid arteries with respect to degree of atherosclerosis and stenosis
Time use of junior doctors performing carotid ultrasound with pocket-sized scanners. | The participants will be followed for the duration of hospital stay, an expected average of approximately 4 days
  Total time used to record the ultrasound images of the carotid arteries by the junior doctors with pocket-sized ultrasound equipment.
Accuracy of high frame rate tracking doppler compared to conventional doppler measurements and computed tomography for grading carotid stenosis. | The participants will be followed for the duration of hospital stay, an expected average of approximately 4 days
  Accuracy of velocity measurements with high frame rate tracking doppler for judging degree of stenosis compared to conventional pulsed wave doppler and computed tomography angiography

OTHER OUTCOMES:
Clinical influence of bed-side ultrasound examinations of the carotid arteries in patients admitted with symptoms of stroke | The participants will be followed for the duration of hospital stay, an expected average of approximately 4 days
  In addition to what described in the primary measure it will be of interest to study predictors of clinical influence of different patient characteristics as age, sex, history, anatomic localization of the vascular event, medication, heart rhythms, ECG findings). Furthermore, the influence on the total cost will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Havard Dalen, MD, PhD, Principal Investigator — Norwegian University of Science and Tehnology
Locations (2):
- Norway (2):
  - Department of Medicine, Hospital of Levanger, Levanger
  - St. Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided
Depending on university's progress for IPD

REFERENCES:
- [Background] Pepi M, Evangelista A, Nihoyannopoulos P, Flachskampf FA, Athanassopoulos G, Colonna P, Habib G, Ringelstein EB, Sicari R, Zamorano JL, Sitges M, Caso P; European Association of Echocardiography. Recommendations for echocardiography use in the diagnosis and management of cardiac sources of embolism: European Association of Echocardiography (EAE) (a registered branch of the ESC). Eur J Echocardiogr. 2010 Jul;11(6):461-76. doi: 10.1093/ejechocard/jeq045. PMID 20702884
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Goldstein LB, Bushnell CD, Adams RJ, Appel LJ, Braun LT, Chaturvedi S, Creager MA, Culebras A, Eckel RH, Hart RG, Hinchey JA, Howard VJ, Jauch EC, Levine SR, Meschia JF, Moore WS, Nixon JV, Pearson TA; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Epidemiology and Prevention; Council for High Blood Pressure Research,; Council on Peripheral Vascular Disease, and Interdisciplinary Council on Quality of Care and Outcomes Research. Guidelines for the primary prevention of stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2011 Feb;42(2):517-84. doi: 10.1161/STR.0b013e3181fcb238. Epub 2010 Dec 2. PMID 21127304
- [Background] Mjolstad OC, Dalen H, Graven T, Kleinau JO, Salvesen O, Haugen BO. Routinely adding ultrasound examinations by pocket-sized ultrasound devices improves inpatient diagnostics in a medical department. Eur J Intern Med. 2012 Mar;23(2):185-91. doi: 10.1016/j.ejim.2011.10.009. Epub 2011 Nov 9. PMID 22284252
- [Background] Skjetne K, Graven T, Haugen BO, Salvesen O, Kleinau JO, Dalen H. Diagnostic influence of cardiovascular screening by pocket-size ultrasound in a cardiac unit. Eur J Echocardiogr. 2011 Oct;12(10):737-43. doi: 10.1093/ejechocard/jer111. Epub 2011 Aug 4. PMID 21821611
- [Background] Fredriksen TD, Avdal J, Ekroll IK, Dahl T, Lovstakken L, Torp H. Investigations of spectral resolution and angle dependency in a 2-D tracking Doppler method. IEEE Trans Ultrason Ferroelectr Freq Control. 2014 Jul;61(7):1161-70. doi: 10.1109/TUFFC.2014.3015. PMID 24960705